CLINICAL TRIAL: NCT01505712
Title: Outcome Prediction in Hodgkin Lymphoma by Low-Density Gene Expression Profiling of Formalin Fixed Paraffin Embedded Tissues: A Correlative Study of Inter-Group Trial E2496
Brief Title: Biomarkers in Tissue Samples From Patients With Hodgkin Lymphoma Enrolled on ECOG-2496 Clinical Trial
Status: Completed | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: CDR0000720334; ECOG-E2496T1
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Lymphoma
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Gene Expression Profiling

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Genetic: gene expression analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors find better ways to treat cancer.

PURPOSE: This research study is studying biomarkers in tissue samples from patients with Hodgkin lymphoma enrolled on ECOG-2496 clinical trial.

DETAILED DESCRIPTION:
OBJECTIVES:

* To explore the predictive power of a gene expression-based multi-gene predictor in classical Hodgkin lymphoma (cHL) with the potential to change clinical practice by basing treatment decisions on biological markers.

OUTLINE: Archived tissue samples are analyzed for gene expression profile using NanoString technology. Results are then compared with patients' treatment outcomes, including failure-free survival and overall survival.

PROJECTED ACCRUAL: A total of 306 patients from ECOG-2496 (training cohort) and 87 patients treated with ABVD in other trials (validation cohort) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Training cohort: Patients diagnosed with locally extensive and advanced stage classical Hodgkin lymphoma (cHL) and treated with doxorubicin, bleomycin, vinblastine, and dacarbazine (ABVD) or mechlorethamine, doxorubicin hydrochloride, vinblastine, vincristine, bleomycin, etoposide, and prednisone (Stanford V)

  * Pretreatment formalin-fixed, paraffin-embedded tissue (FFPET) from patients enrolled on the randomized phase III ECOG-2496 clinical trial
* Validation cohort: Patients with advanced-stage cHL treated with ABVD at the British Columbia Cancer Agency (BCCA)

  * Pretreatment FFPET available

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Samples from patients who participated in E2496 and provided samples for research.
Sampling Method: Non-Probability Sample
Enrollment: 393 (Actual)
Dates: Start 2011-12-15 (Actual); Primary Completion 2012-11-19 (Actual); Study Completion 2012-11-19 (Actual)

PRIMARY OUTCOMES:
Potential of gene expression profiling in changing treatment decision in cHL | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Randall D. Gascoyne, MD, Principal Investigator — British Columbia Cancer Agency